CLINICAL TRIAL: NCT02718469
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of a Monovalent Ebola Zaire Vaccine (rVSVN4CT1-EBOVGP1) Delivered by Intramuscular Injection in Healthy Adult Subjects
Brief Title: Trial to Evaluate Safety and Immunogenicity of an Ebola Zaire Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Auro Vaccines LLC (Industry)
Collaborators: Accelovance (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: rVSV-EBOV-01
Record Dates: First submitted 2016-03-09; First posted 2016-03-24 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Ebola Virus Disease
Keywords: Ebola; VSV; Vesicular Stomatitis Virus; Vaccine; Zaire
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — Ebola Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ebola Vaccine - low dose (Experimental): Low Dose Zaire Ebola Vaccine
  Interventions: Biological: Ebola Vaccine - low dose
- Ebola Vaccine - mid dose (Experimental): Mid Dose Zaire Ebola Vaccine
  Interventions: Biological: Ebola Vaccine - mid dose
- Ebola Vaccine - high dose (Experimental): High Dose Zaire Ebola Vaccine
  Interventions: Biological: Ebola Vaccine - high dose
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Ebola Vaccine - low dose — 2 x 0.5ml vaccine will be given as intramuscular injections on each of day 1 and day 28
  Other Names: Ebola Zaire Vaccine (2.5 x 10^4 pfu)
  Arms: Ebola Vaccine - low dose
Biological: Ebola Vaccine - mid dose — 2 x 0.5ml vaccine will be given as intramuscular injections on each of day 1 and day 28
  Other Names: Ebola Zaire Vaccine (2.5 x 10^5 pfu)
  Arms: Ebola Vaccine - mid dose
Biological: Ebola Vaccine - high dose — 2 x 1.0ml vaccine will be given as intramuscular injections on each of day 1 and day 28
  Other Names: High Dose Ebola Zaire Vaccine (2.0 x 10^6 pfu)
  Arms: Ebola Vaccine - high dose
Biological: Placebo — 2 x 0.5ml or 2 x 1.0ml placebo will be given as intramuscular injections on each of day 1 and day 28 depending on cohort
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety profile of the Zaire Ebola vaccine and the strength of the immune response.

DETAILED DESCRIPTION:
Ebola Zaire is a filovirus that has caused devastating epidemics of hemorrhagic fever in South Africa. Research is underway to create a safe and effective vaccine to protect against Ebola disease, especially for the military and health care workers. Promising animal studies with this vaccine indicate safety and immunogenicity, and the vaccine platform used to deliver the Ebola protein antigen has been successful in creating a safe and protective immune response in people. Note that only one Ebola protein is used in this vaccine; since the entire intact Ebola virus is required for infection, it is impossible to get Ebola disease from this vaccine.

The study targets enrollment of 39 healthy adults. These participants are divided into 3 groups that will be administered one of three dose levels of the vaccine (low, medium, high). The study participants will receive two doses of vaccine: one on day 1 and the second on day 28 (1 month). Three participants at each dose level will act as controls and receive a placebo instead of the active vaccine. A total of 13 visits to the clinic are required over a period of 26 weeks. The total study is expected to take 9 months.

ELIGIBILITY:
INCLUSION CRITERIA:

Subjects who have provided written informed consent and an authorization for disclosure of protected health information must meet the following criteria:

1. Healthy adult men or women, 18 to 60 (inclusive) years of age.
2. Have provided written informed consent prior to screening procedures.
3. Free of clinically significant health problems, as determined by pertinent medical history, physical examination without significant findings in the 28 days prior to enrollment, and clinical judgment of the Investigator.
4. Agrees not to have, or plan to have, non-study vaccines within 60 days after receiving the initial study vaccine, unless medically indicated (i.e., tetanus, rabies vaccine).
5. Agrees not to have contact with ruminant animals or other hoofed animals such as horses, pigs and cows 7 days after each vaccination.
6. Available, able, and willing to participate for all study visits and procedures through Day 182 (Week 26).
7. Be willing to minimize blood and body fluid exposure of others for 7 days after vaccination by:

   * using effective barrier prophylaxis, such as latex condoms, during penetrative sexual intercourse;
   * avoiding the sharing of needles, razors, or toothbrushes; and
   * avoiding open mouth kissing.
8. Body mass index (BMI) less than 40 kg/m2.
9. Laboratory criteria without clinically significant findings within 28 days prior to enrollment:

   * hemoglobin ≥11.5 g/dL for women and ≥13.5 g/dL for men.
   * white blood cell count ≥3500 cells/mm3.
   * differential either within institutional normal range or accompanied by site physician approval;
   * platelets within normal limits;
   * alanine aminotransferase (ALT) or aspartate aminotransferase (AST) and alkaline phosphatase within upper limit of normal range or as approved by the Investigator; and
   * serum creatinine within upper limit of normal range or as approved by the Investigator.
10. Negative for Food and Drug Administration (FDA) approved HIV blood test.
11. Negative hepatitis B surface antigen (HbsAg).
12. Negative antibody to hepatitis C virus (antiHCV).
13. Normal urinalysis defined as negative or trace glucose, protein, and blood (non-menstruating females) by dipstick.
14. Negative urine pregnancy test for women of childbearing potential.
15. Non-pregnant, non-lactating females must meet one of the following criteria: no reproductive potential because of menopause (one year without menses) or because of a hysterectomy, bilateral oophorectomy, or tubal ligation; or subject agrees to be heterosexually inactive at least 21 days prior to enrollment and throughout the duration of the study; or agrees to consistently practice contraception at least 21 days prior to enrollment and throughout the duration of the study by one of the following methods: abstinence, condoms (male or female with or without a spermicide), diaphragm or cervical cap with spermicide, intrauterine device, contraceptive pills or patch, Norplant, Depo-Provera or other FDA approved contraceptive method, or male partner has previously undergone a vasectomy as declared in medical history.

EXCLUSION CRITERIA:

Any subject who meets any of the following criteria will not qualify for entry into the study:

1. History of prior infection with a filovirus or prior participation in a filovirus vaccine trial.
2. History of prior infection with VSV or receipt of a VSV vectored vaccine.
3. Has traveled to an area where the World Health Organization (WHO) has declared as an Ebola outbreak zone.
4. Healthcare worker who has direct contact with patients (nurse, physician, dentist, emergency medical technician, dental hygienist).
5. Has a household contact (HHC) who is immunodeficient, on immunosuppressive medications, HIV positive, pregnant or breast-feeding, or has an unstable medical condition.
6. Breast-feeding, or is a childcare worker, or HHC, who has direct contact with children, 5 years of age or younger.
7. Direct hands-on job preparing food in the food industry.
8. History of employment in an industry involved in contact with ruminant animals, other hoofed animals such as pigs and horses, veterinary sciences, or other potential exposure to VSV.
9. History of employment or activity that involves potential contact with filoviruses.
10. History of severe local or systemic reactions to any vaccination or a history of severe allergic reactions.
11. Known allergy to any rVSVN4CT1 vectored vaccine component.
12. Receipt of investigational product (IP) up to 30 days prior to randomization or ongoing participation in another clinical trial except observational studies.
13. Receipt of licensed non-live or live vaccines within 30 days prior to planned study immunization.
14. Ability to observe possible local reactions at the eligible injection sites (deltoid region) is, in the opinion of the Investigator, unacceptably obscured due to a physical condition or permanent body art.
15. Acute or chronic, clinically significant dermatologic, psychiatric, hematologic, pulmonary, cardiovascular, or hepatic or renal functional abnormality as determined by the Investigator based on medical history, physical examination, and/or laboratory screening test. This would include a known autoimmune arthritis, hemoglobinopathy or coagulation abnormality as judged by the Investigator.
16. Leukopenia due to a clinical or pathological process, unless leukopenia is directly attributable to a transient process (e.g., acute viral infection) and resolution has been documented at time of enrollment.
17. Any screening or baseline laboratory test which in the opinion of the Investigator, is considered clinically significant.
18. Any cytotoxic therapy in the previous 5 years.
19. Diabetes mellitus (type I or II), with the exception of previous gestational diabetes.
20. Any chronic or active neurologic disorder, such as migraines (including silent), seizures or epilepsy (excluding a single febrile seizure as a child as judged by the Investigator).
21. Have a known history of Guillain Barré Syndrome (GBS).
22. Have an active malignancy or history of metastatic or hematologic malignancy.
23. Suspected or known alcohol and/or illicit drug abuse within the past 5 years per the judgment of the Investigator.
24. Moderate or severe illness and/or fever >100.4 °F within 1 week prior to vaccination (subjects can be rescheduled).
25. Administration of immunoglobulin G (IgGs) and/or any blood products within the 120 days preceding study entry or planned administration during the study period.
26. History of blood donation within 60 days of enrollment or plans to donate within the study period.
27. Administration of chronic (defined as more than 14 days) immunosuppressants or other immune modifying drugs within 6 months of study entry: for corticosteroids, this includes chronic oral >14 days or intraarticular steroids in the past 6 months (intranasal and topical are allowed).
28. Major surgery or hospitalization planned during the period of study participation.
29. Research staff or the immediate family of research staff directly involved with the clinical study.
30. Any other significant finding that in the opinion of the Investigator that would increase the risk of the individual having an adverse outcome from participating in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2016-09-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (Safety and Tolerability) | 9 months
  To establish the maximum safe and tolerated dose of a monovalent Ebola Zaire vaccine, as determined by local and systemic reactogenicity signs and symptoms, laboratory measures of safety, and adverse and serious adverse experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Murray A Kimmel, DO, Principal Investigator — Optimal Research, LLC
Locations (1):
- Optimal Research, Melbourne, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clarke DK, Xu R, Matassov D, Latham TE, Ota-Setlik A, Gerardi CS, Luckay A, Witko SE, Hermida L, Higgins T, Tremblay M, Sciotto-Brown S, Chen T, Egan MA, Rusnak JM, Ward LA, Eldridge JH. Safety and immunogenicity of a highly attenuated rVSVN4CT1-EBOVGP1 Ebola virus vaccine: a randomised, double-blind, placebo-controlled, phase 1 clinical trial. Lancet Infect Dis. 2020 Apr;20(4):455-466. doi: 10.1016/S1473-3099(19)30614-0. Epub 2020 Jan 14. PMID 31952923